CLINICAL TRIAL: NCT05099172
Title: An Open Label, First-in-human Study of BAY 2927088 in Participants With Advanced Non-small Cell Lung Cancer (NSCLC) Harboring an EGFR and/or HER2 Mutation
Brief Title: First in Human Study of BAY2927088 in Participants Who Have Advanced Non-small Cell Lung Cancer (NSCLC) With Mutations in the Genes of Epidermal Growth Factor Receptor (EGFR) and/or Human Epidermal Growth Factor Receptor 2 (HER2)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21607; 2023-503795-24-00 (Registry Identifier: CTIS (EU)); 2021-003022-77 (EudraCT Number)
Expanded Access: NCT06761976 (Available)
Record Dates: First submitted 2021-10-19; First posted 2021-10-29 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Advanced Non-small Cell Lung Cancer; EGFR Mutation; HER2 Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose escalation (Experimental): Doses of BAY2927088 will be increased in a stepwise fashion up to the MTD or MAD.
  Interventions: Drug: BAY2927088_formulation A; Drug: BAY2927088_formulation B_1; Drug: BAY2927088_formulation B_2
- Backfill (Experimental): Dose Escalation and Backfill run concurrently
  Interventions: Drug: BAY2927088_formulation A; Drug: BAY2927088_formulation B_1; Drug: BAY2927088_formulation B_2
- Dose expansion (Experimental): Eight independent groups (group A, B1, B2, C, D, E, F, G) are planned. Dose Expansion may start at a dose level that has been evaluated in Escalation/Backfill in at least 9 participants and considered safe or at any other dose levels that are below the highest dose level that is considered safe.
  Interventions: Drug: BAY2927088_formulation B_1; Drug: BAY2927088_formulation B_2
- Extension part (Experimental): Initiation of the Extension part will depend on the benefit-risk profile observed during Dose Expansion. Additionally, enrollment may be prematurely terminated based on emerging data at the discretion of the Sponsor.
  Interventions: Drug: BAY2927088_formulation B_1; Drug: BAY2927088_formulation B_2

INTERVENTIONS:
Drug: BAY2927088_formulation A — Oral administration
  Arms: Backfill; Dose escalation
Drug: BAY2927088_formulation B_1 — Oral administration
Drug: BAY2927088_formulation B_2 — Oral administration

SUMMARY:
Researchers are looking for a better way to treat people who have advanced non-small cell lung cancer (NSCLC), a group of lung cancers that have spread to nearby tissues or to other parts of the body.

Epidermal growth factor receptor (EGFR) and human epidermal growth factor receptor 2 (HER2) are proteins that help cells to grow and divide. A damage (also called mutation) to the building plans (genes) for these proteins in cancer cells leads to a production of abnormal EGFR and/or HER2. These abnormal proteins drive the growth and the spread of the cancer. Several EGFR and/or HER2 mutations exist in the cancer cells. The study treatment, BAY2927088, is expected to block the mutated EGFR and HER2 proteins which may stop the spread of NSCLC.

The main purpose of this study is to learn:

Escalation, Backfill, and Expansion Part:

* How safe is BAY2927088 for the participants?
* What is the highest dose of BAY2927088 that can be tolerated (maximum tolerated dose) by or given to (maximum administered dose) the participants?
* How does BAY2927088 move into, through, and out of the bodies of the participants?

For this, the researchers will measure the followings:

* The number of participants with medical problems, also called adverse events and serious adverse events, and their severity
* The number of participants who discontinue study treatment due to an adverse event.
* The highest dose of BAY2927088 that the participants can take without having adverse events (maximum tolerated dose (MTD)) or the maximum dose that is tested and found to be safe for the participants in case MTD cannot be found out (maximum administered dose (MAD)) of BAY2927088
* Number of participants experiencing adverse events that prevent an increase in the dose of BAY2927088 (dose-limiting toxicities (DLTs)) at each dose level
* The (average) total level of BAY2927088 in the blood (also called AUC) after receiving single or multiple doses of BAY2927088
* The (average) highest level of BAY2927088 in the blood (also called Cmax) after receiving a single or multiple doses of BAY2927088 Extension Part
* How well does BAY2927088 work in participants?

For this, the researchers will measure the following:

• Percentage of participants whose cancer completely disappears (complete response) or reduces by at least 30% (partial response) after taking the treatment (also known as objective response rate (ORR)). This will be assessed by doctors other than the study doctor.

This study has 4 parts:

* The escalation part aims to find the maximum daily amount (dose) of BAY2927088 that participants can receive.
* The backfill part aims to test the doses of BAY2927088 that are considered safe in the escalation part by giving it to more participants. This will help find optimal doses of BAY2927088 that work well and are safe to be tested in the next part.
* The expansion part aims to determine the dose of BAY2927088 to be tested in further studies.
* The extension part aims to determine whether the selected dose of BAY2927088 from the expansion part works well.

The participants in this study will take the study treatment BAY2927088 in 3-week periods called "cycles". They will in general take BAY2927088 once or twice daily as a liquid/tablet by mouth until their cancer gets worse, they have medical problems, they leave the study, or the study is terminated. Participants will have no more than 5 visits per cycle.

During the study, the study team will:

* take blood and urine samples,
* check the status of the cancer by doing computed tomography (CT) or magnetic resonance imaging (MRI) scans,
* check the participants' overall health and heart health,
* ask the participants questions about how they are feeling and what adverse events they are having.

An adverse event is considered "serious" when it leads to death, puts the participant's life at risk, requires hospitalization, causes disability, causes a baby being born with medical problems, or is medically important.

ELIGIBILITY:
Inclusion Criteria:

* Documented histologically or cytologically confirmed locally advanced NSCLC, not suitable for definitive therapy or recurrent or metastatic NSCLC at screening (small cell or mixed histologies are excluded).
* Documented disease progression after treatment with at least one prior systemic therapy for advanced disease. Participants who do not have standard of care access due to any reason, are intolerant to, or are not eligible for standard treatments, may also be eligible.

Note: Except for participants eligible for one of the groups (Expansion or Extension) who should have received no prior systemic treatment for locally advanced or metastatic disease.

* Adequate archival tumor tissue (ideally taken after last targeted treatment and not older than 6 months) has to be available, either from primary or metastatic sites. If archival material is not available, a fresh tumor biopsy should be performed if feasible and if the procedure poses no significant risk for the participant.
* Measurable disease by RECIST v1.1 with at least one lesion not chosen for biopsy during the screening period (if a biopsy is taken during screening) that can be accurately measured at baseline with computed tomography (CT) or magnetic resonance imaging (MRI) and that is suitable for accurate repeated measurements. A biopsied lesion should not be used as a target lesion for RECIST 1.1 tumor assessments (or, for participants in Expansion Group G, for RANO-BM tumor assessments). Previously irradiated lesions must have shown progression to be considered measurable.
* Documented activating EGFR and/or HER2 mutation assessed by a Clinical Laboratory Improvement Amendments (CLIA)-certified (United States [US] sites) or an equally accredited (outside of the US) local laboratory
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Minimum life expectancy of 12 weeks.
* Adequate bone marrow function as assessed by the following laboratory tests to be conducted within 7 days before the first dose of study treatment:

  1. Hemoglobin ≥ 9.0 g/dL. Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within 2 weeks prior to testing.
  2. Platelets ≥ 100 × 10^9 cells/L.
  3. Absolute neutrophil count ≥ 1.5 ×10^9 cells/L. Criteria must be met without the use of hematopoietic growth factors (e.g., G-CSF) within 2 weeks prior to testing.
* Adequate kidney function as assessed by following laboratory test to be conducted within 7 days before the first dose of study treatment:

  a. Estimated glomerular filtration rate (eGFR) > 50 mL/min per 1.73 m^2 according to the Modification of Diet in renal Disease Study Group (MDRD) formula.
* Adequate liver function as assessed by following laboratory tests to be conducted within 7 days before the first dose of study treatment:

  1. Total bilirubin ≤ 1.5 × ULN (or ≤ 3 X ULN for participants with documented Gilbert-Meulengracht Syndrome, or for participants with hyperbilirubinemia considered due to liver metastasis).
  2. Aspartate transaminase and alanine transaminase ≤ 2.5 × ULN (or ≤ 5 × ULN if due to liver involvement by tumor).

Exclusion Criteria:

* Treatment with an EGFR tyrosine kinase inhibitor (TKI) ≤ 8 days or 5x the terminal phase, elimination half-lives, whichever is shorter, prior to the first dose of study drug.
* Treatment with a systemic anti-cancer treatment (excluding EGFR TKIs as described above) ≤ 14 days prior to the first dose of study drug.
* Radiation therapy, stereotactic radiosurgery (SRS) and palliative radiation ≤ 14 days prior to the first dose of study drug.
* Treatment with immunotherapy ≤ 28 days prior to the first dose of study drug.
* Have any unresolved toxicity of Grade ≥ 2 from previous anti-cancer treatment, except for alopecia and skin pigmentation. Participants with chronic, but stable Grade 2 toxicities may be allowed to enroll after agreement between the Investigator and Sponsor.
* Any history of primary brain or leptomeningeal disease (symptomatic or asymptomatic), presence of symptomatic central nervous system (CNS) metastases, or CNS metastases that require local treatment (such as radiotherapy or surgery).
* History of spinal cord compression or brain metastases with the following exceptions:

  1. Participants with treated brain metastases that are asymptomatic at screening and who are off or receiving low-dose corticosteroids (≤10 mg prednisone or equivalent) for at least 7 days prior to first dose of BAY 2927088 are eligible to enroll in Dose Escalation and Backfill.
  2. Participants with treated brain metastases that are asymptomatic at screening are eligible in Dose Expansion/Extension (with the exception of Group G) if all of the following criteria are met:

     * there is no evidence of progression (new or enlarging brain metastases) for at least 4 weeks after CNS-directed treatment, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period.
     * Participants must be off or receiving low-dose corticosteroids (≤10 mg prednisone or equivalent) for 7 days prior to first dose of BAY2927088.
  3. Participants with history of spinal cord compression >3 months from definitive therapy and stable by imaging (MRI or CT) during the screening period and clinically asymptomatic.
  4. Expansion Group G only: Participants with active (new or progressing) clinically stable brain metastases who do not require immediate CNS-directed treatment as per Investigator's judgement and who are off or receiving low-dose corticosteroids (≤10 mg prednisone or equivalent such as ≤ 1.5 mg/day dexamethasone) in the 7 days prior to first dose of BAY2927088 are eligible.
* History of congestive heart failure (CHF) Class >II according to the New York Heart Association (NYHA) Functional Classification or serious cardiac arrhythmias requiring treatment (e.g. ventricular arrhythmias, atrial fibrillation) or any clinically important abnormalities in rhythm, conduction or morphology or resting ECG (e.g., complete left bundle branch block, third degree heart block, second degree heart block, PR interval >250 msec)
* Participants with:

  1. Known human immunodeficiency virus (HIV), except as noted below: Participants with history of HIV infection are eligible at the Investigator's discretion provided that: • CD4+ T-cell (CD4+) counts are ≥ 350 cells/uL • The participant has been on established antiretroviral therapy (ART) for at least 4 weeks prior to the start of study drug and has an HIV viral load less than 400 copies/mL prior to start of the study treatment • The ART being used does not contain strong inducers or inhibitors of CYP3A4, and is not anticipated to cause overlapping toxicities with study drug • The participant has not had an opportunistic infection within the past 12 months
  2. Active Hepatitis B infection (positive for Hepatitis B surface antigen [HbsAg]) and Hepatitis B virus [HBV] DNA).
  3. Active Hepatitis C infection (positive anti-HCV Antibody and quantitative HCV RNA results greater than the lower limits of detection of the assay).

     NOTE: Participants with history of chronic HBV or HCV infection are eligible at the Investigator's discretion provided that the disease is stable and sufficiently controlled under treatment.
* Use of strong CYP3A4 inhibitors and inducers from 14 days prior to first administration of study drug. Strong CYP3A4 inhibitors and inducers are prohibited during the study and until Safety FU (follow up) visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Up to 30 days after the last administration of study treatment
Number of participants with treatment-emergent serious adverse events (TESAEs) | Up to 30 days after the last administration of study treatment
Severity of TEAEs | Up to 30 days after the last administration of study treatment
Severity of TESAEs | Up to 30 days after the last administration of study treatment
Number of participants who discontinue study treatment due to an AE | About 4 years (Up to the end of study treatment)
Maximum tolerated dose (MTD) or maximum administered dose (MAD) of BAY2927088 within the DLT observation period in Dose Escalation (including participants from Backfill qualifying for the MTD population) | At the end of Cycle 1 of a 21-day cycle
Number of participants experiencing dose-limiting toxicities (DLTs) at each dose level associated with administration of BAY2927088 in the DLT observation period in Dose Escalation (including participants from Backfill) | At the end of Cycle 1 of a 21-day cycle
  In Dose Escalation (including participants from Backfill)
Cmax of BAY2927088 | Cycle 1, Day 1 (Cycle duration is 21 days)
  Cmax: Maximum/peak concentration
AUC(0-24) of BAY2927088 for QD | Cycle 1, Day 1 (Cycle duration is 21 days)
  AUC: Area under the concentration vs. time curve. AUC(0-24): AUC from time 0 to 24 hours post dose. QD: Quaque die (once daily)
AUC(0-12) of BAY2927088 for BID | Cycle 1, Day 1 (Cycle duration is 21 days)
  If applicable. AUC(0-12): AUC from time 0 to 12 hours post dose. BID: Bis in die, 2 times daily.
Cmax,md of BAY2927088 | Cycle 1, Day 15 (Cycle duration is 21 days)
  Cmax,md: Cmax after multiple dose administrations
AUC(0-24)md of BAY2927088 for QD | Cycle 1, Day 15 (Cycle duration is 21 days)
  AUC(0-24)md: AUC(0-24) after multiple dose administrations
AUC(0-12)md of BAY2927088 for BID | Cycle 1, Day 15 (Cycle duration is 21 days)
  If applicable AUC(0-12)md: AUC(0-12) after multiple dose administrations
Overall response rate (ORR) per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1) by blinded independent central review (BICR) in extension part | From the start of the study treatment up to 12 months

SECONDARY OUTCOMES:
Overall response rate (ORR) as per RECIST v1.1 by investigator assessment | About 4 years
  RECIST v1.1: Response Evaluation Criteria in Solid Tumors, version 1.1
Recommended phase 2 dose (RP2D) of BAY2927088 | About 1.5 years
ORR per RECIST v1.1 by Investigator assessment in extension part | From the start of the study treatment up to 12 months
Disease control rate (DCR) per RECIST v1.1 by Investigator assessment and BICR in extension part | From the start of the study treatment up to 12 months
Duration of response (DOR) per RECIST 1.1 by Investigator assessment and BICR in extension part | From the start of the study treatment up to 12 months
Progression-free survival (PFS) per RECIST 1.1 by Investigator assessment and BICR in extension part | From the start of the study treatment up to 12 months
Overall survival (OS) in extension part | From the start of the study treatment up to 12 months
Number of participants with treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events (TESAEs) categorized by severity in extension part | Up to 30 days after the last administration of study treatment

CONTACTS AND LOCATIONS:
Locations (81):
- United States (10):
  - Banner MD Anderson Cancer Center at Banner Gateway Medical Center, Gilbert, Arizona
  - City of Hope - Duarte Cancer Center, Duarte, California
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - The Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Dana-Farber Cancer Institute - Oncology Department, Boston, Massachusetts
  - Brigette Harris Cancer Pavilion at Henry Ford Cancer Center - Detroit, Detroit, Michigan
  - NYU Langone Hospital - Long Island - Urology, Mineola, New York
  - Tennessee Oncology - Nashville Centennial Clinic, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center - Texas Medical Center, Houston, Texas
  - Virginia Cancer Specialists, PC - Fairfax, Fairfax, Washington
- Belgium (2):
  - UZ Leuven Gasthuisberg - Pneumology Department, Leuven, Vlaams-Brabant
  - AZ Delta | Clinical Trial Center - Pneumology, Roeselare, West-Flanders
- Brazil (2):
  - Liga Norte Riograndense Contra o Cancer | Centro de Pesquisa Clínica, Natal, Rio Grande do Norte
  - Hospital de Base | Integrated Research Center, São José do Rio Preto, São Paulo
- China (14):
  - Beijing Cancer Hospital - Oncology Department, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Union Hospi, Tongji Med College, Huazhong Univ. Scien&Tech, Wuhan, Hubei
  - Hunan Cancer Hospital - Oncology Department, Changsha, Hunan
  - NJ Drum Tower Hospital, the Affil Hos of NJ Univ Med School, Nanjing, Jiangsu
  - Qilu Hosp., Shandong Univ., Jinan, Shandong
  - Shandong University - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai Chest Hospital, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital, Zhejiang Univ. School of Medicine - Oncology Department, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang University School of Medicine - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
- France (6):
  - Institut Bergonie - Unicancer Nouvelle Aquitaine - Service Oncologie medicale, Bordeaux
  - UNICANCER - Centre Leon-Berard (CLB) - Medical oncology, Lyon
  - Hopital Nord Laennec - Oncologie medicale thoracique et digestive, Nantes
  - Institut Curie - Paris - Oncologie medicale, Paris
  - Institut de Cancerologie Ouest - Saint Herblain - Oncologie medicale, Saint-Herblain
  - Gustave Roussy - Departement Oncologie-Radiotherapie, Villejuif
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong, Hong Kong SAR
  - Queen Mary Hospital, Hong Kong, Hong Kong SAR
- Israel (2):
  - Rabin Medical Center | Beilinson Hospital - Internal Medicine C Department, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
- Italy (8):
  - Azienda Ospedaliero Universitaria Parma - SC Oncologia Medica, Parma, Emilia-Romagna
  - Centro di Riferimento Oncologico di Aviano - Oncologia Medica e dei Tumori Immuno-Correlati, Aviano, Friuli Venezia Giulia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOC Fase I, Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori - S. C. Oncologia Medica 1, Milan, Lombardy
  - Istituto Europeo di Oncologia s.r.l - Sviluppo di nuovi farmaci per Terapie Innovative, Milan, Lombardy
  - Humanitas Mirasole S.p.A. - Oncologia Medica ed Ematologia, Rozzano, Lombardy
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga - Oncologia Medica, Orbassano, Piedmont
  - Centro Ricerche Cliniche Di Verona S.r.l. - Oncologia, Verona
- Japan (11):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Sakai, Osaka
  - Shizuoka Cancer Center, Sunto, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Tottori University Hospital, Yonago, Tottori
  - Okayama University Hospital, Okayama
- Netherlands (2):
  - Nederlands Kanker Instituut, Amsterdam
  - Erasmus University Medical Center | Research Department - Lung Diseases, Rotterdam
- IPO Porto, Porto, Portugal
- Singapore (3):
  - National University Hospital Medical Centre, Singapore
  - National Cancer Center Singapore - Oncology Department, Singapore
  - Curie Oncology | Mount Elizabeth Novena, Singapore
- South Korea (7):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - St.Vincent's Hospital, Suwon, Gyeonggido
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Severance Hospital, Yonsei University Health System - Oncology Department, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center | Oncology, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center - Oncology Department, Seoul
- Spain (6):
  - Institut Catala D'oncologia | Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Dexeus Grupo Quironsalud | Oncologia, Barcelona
  - Hospital Universitari Vall D Hebron | Oncologia, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz | Oncologia, Madrid
  - Hospital Universitario Hm Sanchinarro | Oncologia, Madrid
  - Hospital Universitario Y Politecnico La Fe | Oncologia, Valencia
- Taiwan (5):
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi-Mei Medical Center, Liouyine, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital at Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Le X, Kim TM, Loong HH, Prelaj A, Goh BC, Li L, Fang Y, Lu S, Dong X, Wu L, Shinno Y, Daniele G, Yang TY, Kim HR, Ruiter G, Zhao J, Novello S, Miao L, Janne PA, Goto K, Ruttinger D, Descamps T, Brase JC, Bao W, Li R, Brega N, Grassi P, Girard N, Tan DS; SOHO-01 Investigators. Sevabertinib in Advanced HER2-Mutant Non-Small-Cell Lung Cancer. N Engl J Med. 2025 Nov 6;393(18):1819-1832. doi: 10.1056/NEJMoa2511065. Epub 2025 Oct 17. PMID 41104928